CLINICAL TRIAL: NCT01263574
Title: Trial of Ethanol Lock Therapy to Prevent Catheter Associated Blood Stream Infections
Brief Title: Trial of 70% Ethanol Versus Heparin to Reduce the Rate of Central Line Infections in Children With Short Bowel Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants. IND denied by FDA.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Tom Jaksic, W. Hardy Hendren Professor of Surgery, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-03-0132
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Catheter Related Infections; Short Bowel Syndrome
Keywords: Catheter related infections prevention/control; Anti infective agents; Catheter related infections prevention
MeSH Terms: conditions — Catheter-Related Infections; Short Bowel Syndrome | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparinized Saline (Placebo Comparator): This group will maintain their central lines patent with heparinized saline.
  Interventions: Drug: 70% ethanol
- Ethanol lock solution group (Experimental): Administration of the 70% ethanol lock solution will occur between cycles of parenteral nutrition. Randomized lock solutions will be administered three days per week. When patients have completed their parenteral nutrition, their central venous catheters will be flushed with 5mL saline, per current standards
  Interventions: Drug: 70% ethanol

INTERVENTIONS:
Drug: 70% ethanol — Administration of the lock solution will occur between cycles of parenteral nutrition. Lock solutions will be administered three days per week. The pre-measured volume of lock solution will then be injected into the catheter for 4 hours. Prior to the next instillation of medications into the catheter, the lock solution will be aspirated and discarded. Another 5mL flush of saline will then be instilled into the catheter prior to medication or parenteral nutrition administration. Volume of lock solution administered will be determined by catheter size.
  Other Names: ethanol lock

SUMMARY:
This study is designed to determine if the use of 70% ethanol lock solution in central lines decreases the rate of central line infections in children with short bowel syndrome. While ethanol locks have been used safely in children, there has been no published research to date that clearly shows it is of definite benefit in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >3 months
* Intestinal failure patients
* Silicone catheter for the administration of parenteral nutrition

Exclusion Criteria:

* Age < 3 months
* Weight < 5 kg
* Documented allergy to ethanol
* Evidence of tunnel site infection
* Patients receiving continuous renal replacement therapy
* Concomitant use of metronidazole

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02 (Estimated); Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Catheter associated blood stream infection (CABSI). | Number of infections reported per 1000 catheter days.
  Published data in intensive care unit (ICU) patients with CABSI has noted that central venous catheter cultures had a specificity of 98% and a negative predictive value of 97%. In our study, we will define CABSI as a positive central venous catheter blood culture in the face of clinical signs of infection, when the catheter has been used in the last 48 hours prior to infection, and without other obvious source of infection. CABSI rate will be reported as number of infections per 1000 catheter days after 12 months of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Jaksic, M.D, Ph.D, Principal Investigator — Boston Children's Hospital; Christopher Duggan, M.D, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No